CLINICAL TRIAL: NCT03708744
Title: A Randomized Open-label 4-way Crossover Study to Compare the PK, Safety, and Tolerability of M207 at Two Different Application Locations for 30 Minutes With Intranasal Zolmitriptan 2.5 mg and 1 Hour Wear Time in Healthy Volunteers
Brief Title: A Study of M207 With Intranasal Zolmitriptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-2018-002
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Migraine
Keywords: Healthy; Volunteer; Pharmacokinetics
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, open-label four-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Treatment A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application)
  Interventions: Drug: A: M207 3.8mg, 30 min, upper arm; Drug: B: M207 3.8 mg, 30 min, thigh; Drug: C: M207 3.8 mg, 1 hr, upper arm; Drug: D:zolmitriptan nasal spray
- Treatment B (Experimental): Treatment B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application)
  Interventions: Drug: A: M207 3.8mg, 30 min, upper arm; Drug: B: M207 3.8 mg, 30 min, thigh; Drug: C: M207 3.8 mg, 1 hr, upper arm; Drug: D:zolmitriptan nasal spray
- Treatment C (Experimental): Treatment C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application)
  Interventions: Drug: A: M207 3.8mg, 30 min, upper arm; Drug: B: M207 3.8 mg, 30 min, thigh; Drug: C: M207 3.8 mg, 1 hr, upper arm; Drug: D:zolmitriptan nasal spray
- Treatment D (Active Comparator): Treatment D: Intranasal zolmitriptan 2.5 mg
  Interventions: Drug: A: M207 3.8mg, 30 min, upper arm; Drug: B: M207 3.8 mg, 30 min, thigh; Drug: C: M207 3.8 mg, 1 hr, upper arm; Drug: D:zolmitriptan nasal spray

INTERVENTIONS:
Drug: A: M207 3.8mg, 30 min, upper arm — A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application)
  Other Names: A: Zolmitriptan patch, 3.8 mg, 30 min, upper arm
Drug: B: M207 3.8 mg, 30 min, thigh — B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application)
  Other Names: B: Zolmitriptan patch 3.8 mg, 30 min, thigh
Drug: C: M207 3.8 mg, 1 hr, upper arm — C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application)
  Other Names: C: Zolmitriptan patch, 3.8 mg, 1 hour, upper arm
Drug: D:zolmitriptan nasal spray — D: 2.5 mg/0.1 mL intranasal zolmitriptan
  Other Names: Zomig Nasal Spray

SUMMARY:
This is a single-center, open-label, randomized, four-way crossover study. Each subject will receive each of the four study treatments once, followed by in-clinic monitoring and extensive blood sample collection for pharmacokinetic analysis.

Dosing will occur approximately 48 hours apart, until completion of dosing in randomized order per the treatment sequence tables. Plasma samples from the dosing days will be sent to the analytical laboratory for analysis and tolerability for each of the dose levels will be summarized.

After completion of the four dosing days, subjects will be assessed one final time and dismissed from the study.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, four-way crossover study to compare the pharmacokinetics, safety and tolerability of:

M207 3.8 mg administered to the upper arm to M207 3.8 mg administered to the thigh, particularly with respect to skin irritation (erythema, edema, bruising, bleeding):

M207 3.8 mg worn for 30 minutes on the upper arm to M207 3.8 mg worn for 1 hour on the upper arm; and M207 3.8 mg to intranasal zolmitriptan 2.5 mg.

Each subject will receive each of the four study treatments once, followed by in-clinic monitoring and extensive blood sample collection for pharmacokinetic analysis.

M207 application sites will be observed for erythema, edema, bruising, and bleeding at various timepoints throughout the study.

Dosing will occur approximately 48 hours apart, until completion of dosing in randomized order per the treatment sequence tables. Plasma samples from the dosing days will be sent to the analytical laboratory for analysis and tolerability for each of the dose levels will be summarized.

After completion of the four dosing days, subjects will be assessed one final time and dismissed from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men 18 to 50 years of age.
2. Good general health with no clinically significant abnormalities as determined by medical history, physical examination, complete blood count (CBC), blood chemistry, urinalysis, and ECG.
3. Negative urine drug and alcohol screens and negative serum pregnancy tests (for female subjects) at screening.
4. Consent of female subjects to use a medically effective method of contraception throughout the entire study period and for 30 days after the subject completes the study. Medically effective methods of contraception that may be used by the subject include abstinence, use of diaphragm and spermicide, intrauterine device (IUD), condom and vaginal spermicide, hormonal contraceptives (subjects must be stable on hormonal contraceptives for at least the prior 3 months), surgical sterilization, and post-menopausal (≥ 2 years of amenorrhea).
5. Ability to read, understand, and provide written informed consent that they understand the purpose of the study and procedures required for the study before enrolling in the study, and willingness to comply with all study procedures and restrictions.

Exclusion Criteria:

1. Evidence of significant history of hepatic, reproductive, gastrointestinal, renal, bleeding, or hematological disorders including coagulation, pulmonary, neurological, respiratory, endocrine, or cardiovascular system abnormalities (especially hypertension, peripheral vascular disease, coronary artery disease, transient ischemic attacks, or cardiac rhythm abnormalities), psychiatric disorders, acute infection, or other conditions that would interfere with study participation or with the absorption, distribution, metabolism, or excretion of drugs.
2. Presence of two or more risk factors for cardiovascular disease (family history of premature heart disease, hyperlipidemia, or hypertension)
3. Any contraindication to zolmitriptan administration including:

   * History of coronary artery disease or coronary vasospasm
   * Symptomatic Wolf-Parkinson-White syndrome or other cardiac accessory conduction pathway disorders
   * History of stroke, transient ischemic attack, or hemiplegic or basilar migraine
   * Peripheral Vascular Disease
   * Ischemic bowel disease
   * Uncontrolled hypertension
   * Any history of hepatic impairment
4. History of contact dermatitis or known dermatological disorders that would interfere with the study procedures or assessments
5. Planned participation in activities which cause inflammation, irritation, sunburn, lesions, or tattoos at the intended application sites from 2 weeks prior to screening through their last day of study participation
6. Use of warfarin within 1 month prior to the first dose or heparin within 1 week prior to study drug administration
7. Use of prescription and over the counter medications other than the following:

   * Hormone Replacement Therapy (HRT)
   * Birth control pills, patches, injections, or implants (all hormonal contraceptives) are allowed provided the dose has been stable for at least one month prior to screening and may be continued throughout the study
   * Antihistamines
   * Intermittently used NSAIDS
   * Acetaminophen if medically necessary (not more than 2 g/day)
   * Exceptions may be allowed on a case by case basis
8. Subjects who have a known allergy or sensitivity to zolmitriptan or its derivatives or formulations
9. Known allergy or sensitivity to tapes, adhesives, or zolmitriptan
10. Regular or recent intake of prescription drugs, particularly drugs with an influence on blood pressure.
11. Use of any other investigational compound within one month of planned study drug dosing
12. On-going drug or alcohol abuse, or history of either deemed to be clinically significant by the investigator
13. Systolic BP (measured after remaining sitting for 5 minutes) greater than 140 mmHg and diastolic BP greater than 90 mmHg at screening
14. History of nasal pathology (e.g., polyps) or abnormal nasal exam
15. Body Mass Index (BMI) greater than 35 kg/m2
16. If, in the opinion of the investigator, the subject is not suitable for the study
17. Any positive urine drug screen result or alcohol breath test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Kellerman, Pharm.D., Study Director — Zosano Pharma Corporation
Locations (1):
- Hill Top Research, Inc., Neptune City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4-way crossover, each subject randomized to receive A, B, C, and D in one of four sequences.
  A: M207 3.8 mg, two 1.9 mg patches, 30 min, upper arm B: M207 3.8 mg, two 1.9 mg patches, 30 min, thigh C: M207 3.8 mg, two 1.9 mg patches, 1 hr, upper arm D: Intranasal zolmitriptan 2.5 mg One subject randomized to CADB was given ABCD.
Groups:
- ABCD: A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application) B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application) C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application) D: Intranasal zolmitriptan 2.5 mg
- BDAC: B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application) D: Intranasal zolmitriptan 2.5 mg A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application) C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application)
- CADB: C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application) A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application) D: Intranasal zolmitriptan 2.5 mg B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application)
- DCBA: D: Intranasal zolmitriptan 2.5 mg C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application) B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application) A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application)
Period: Overall Study
Arm/Group | ABCD | BDAC | CADB | DCBA
Started | 7 | 6 | 5 | 6
Completed | 7 | 6 | 4 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Each subject received each of the four treatments below in one of four treatment sequences.
  A: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (upper arm application) B: M207 3.8 mg administered as two 1.9 mg patches, 30 min wear time (thigh application) C: M207 3.8 mg administered as two 1.9 mg patches, 1 hour wear time (upper arm application) D: Intranasal zolmitriptan 2.5 mg
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.93 (3.264)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: maximum observed plasma concentration
Time Frame: pre-dose, 2, 5, 10, 15, 20, 30, 45, 60, 90 minutes, 2, 4, 8, 12, 24 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 22 | 23 | 23
pg/mL | 9180.9 (4066.1) | 5925.9 (2353.3) | 15224.3 (12972.9) | 3758.3 (1711.6)

2. Secondary Outcome: Adverse Events
Description: number of subjects that experienced at least one adverse event
Time Frame: 24 hours
Population: Subjects who received treatment
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23 | 24 | 23
Participants | 4 | 3 | 1 | 1

3. Secondary Outcome: t(1/2)
Description: apparent half-life
Time Frame: pre-dose, 2, 5, 10, 15, 20, 30, 45, 60, 90 minutes, 2, 4, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 21 | 23 | 19
hours | 2.692 (0.486) | 2.975 (1.217) | 2.959 (0.998) | 4.545 (1.535)

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 4/23 | 3/23 | 1/24 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=23) | Treatment B (N=23) | Treatment C (N=24) | Treatment D (N=23)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intranasal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03708744/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03708744/SAP_001.pdf